CLINICAL TRIAL: NCT02266485
Title: Pharmacodynamics, Preliminary Pharmacokinetics and Tolerability After Multiple Oral Doses of 2.5 mg o.d. BIBB 515 BS (Capsule) or Pravastatin 20 mg Over 2 Weeks in Hyperlipemic Healthy Male Subjects (Parallel Group Comparison, Randomized, Placebo Controlled, Partly Double Blind [Pravastatin Open])
Brief Title: Pharmacodynamics, Preliminary Pharmacokinetics and Tolerability of BIBB 515 BS or Pravastatin in Hyperlipemic Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 525.3
Record Dates: First submitted 2014-10-16; First posted 2014-10-17 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Pravastatin

ARMS (3):
- BIBB 515 BS (Experimental)
  Interventions: Drug: BIBB 515 BS
- Pravastatin (Active Comparator)
  Interventions: Drug: Pravastatin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIBB 515 BS
  Arms: BIBB 515 BS
Drug: Pravastatin
  Arms: Pravastatin
Drug: Placebo
  Arms: Placebo

SUMMARY:
Investigation of pharmacodynamics (inhibition of oxidosqualene cyclase, MES as marker), effect on routine lipid profile parameters, safety and preliminary pharmacokinetics

ELIGIBILITY:
Inclusion Criteria:

* Healthy male caucasian subjects as determined by results of screening
* Written informed consent in accordance with good clinical practice (GCP) and local legislation given
* Age ≥ 18 and ≤ 65 years
* Broca ≥ - 20 % and ≤ + 30 %
* Cholesterol level ≥ 5.4 mmol/l

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurologic disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which was deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) (≤ 1 month prior to administration or during the trial)
* Use of any drugs which might influence the results of the trial (≤ 10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (≤ 2 months prior to administration or during the trial)
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day)
* Inability to refrain from smoking on study days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation > 100 ml (≤ 4 weeks prior to administration or during the trial)
* Excessive physical activities (≤ 10 days prior to administration or during the trial)
* Any laboratory value outside the reference range of clinical relevance
* Abnormal findings at eye lens examination

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 1998-07; Primary Completion 1998-09 (Actual)

PRIMARY OUTCOMES:
Percentage changes in total-cholesterol | Pre-dose, up to day 15
Percentage changes in low density lipoprotein (LDL) - cholesterol | Pre-dose, up to day 15
Percentage changes in high density lipoprotein (HDL) - cholesterol | Pre-dose, up to day 15
Percentage changes in apo-lipoprotein B | Pre-dose, up to day 15
Percentage changes in lipoprotein (a) | Pre-dose, up to day 15
Percentage changes in triglycerides | Pre-dose, up to day 15
Maximum concentration of the analyte in plasma at different time points (Cmax) | Up 336 hours after first drug administration
Time to reach maximum concentration of the analyte in plasma at different time points (tmax) | Up 336 hours after first drug administration
Apparent terminal elimination half-life of the analyte in plasma (t1/2) | Up 336 hours after first drug administration
Area under the concentration-time curve of the analyte in plasma at different time points (AUC) | Up 336 hours after first drug administration
Total mean residence time of the analyte in the body (MRTtot) | Up 336 hours after first drug administration
Apparent clearance of the analyte in plasma after extravascular multiple dose administration (CL/f) | Up 336 hours after first drug administration
Apparent volume of distribution of the analyte during the terminal phase (Vz/f) | Up 336 hours after first drug administration
Terminal rate constant of the analyte in plasma (λz) | Up 336 hours after first drug administration
Number of participants with clinically relevant changes from baseline in physical examination | Pre-dose and day 15
Number of participants with clinically relevant changes from baseline in 12-lead ECG | Pre-dose and day 15
Number of participants with clinically relevant changes from baseline in lens examination | Pre-dose and day 15
Number of participants with clinically relevant changes in vital signs (blood pressure, pulse rate, body weight) | Pre-dose, up to 324 hours after first drug administration
Number of participants with clinically relevant changes in laboratory parameters | Pre-dose, up to 324 hours after first drug administration
Number of participants with adverse events | Up to 1 day after last drug administration
Global clinical assessment by the investigator | On day 15 after first drug administration
Monoepoxy-squalene (MES) plasma concentration at different time points | Pre-dose, up to day 15
  as surrogate marker for squalene inhibition